CLINICAL TRIAL: NCT02766478
Title: Genistein Supplementation to Mitigate Cardiometabolic Dysfunction in Patients Undergoing Androgen Deprivation Therapy for Prostate Cancer
Acronym: GeniPro
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment and study activities were suspended due to COVID-19.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jessica Alvarez, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00086186
Record Dates: First submitted 2016-05-06; First posted 2016-05-09 (Estimated); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Genistein (Experimental): Participants with and without diabetes will receive 60 mg/day oral genistein (30 mg taken twice daily) for 12 weeks.
  Interventions: Drug: Genistein
- Placebo (Placebo Comparator): Participants with and without diabetes will receive placebo taken twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Genistein — Genistein is a natural supplement that comes from soy. Genistein will be taken orally (30 mg twice daily) for 12 weeks.
  Arms: Genistein
Drug: Placebo — A placebo pill will be taken orally for 12 weeks.
  Arms: Placebo

SUMMARY:
Genistein is a natural supplement that comes from soy. The purpose of this study is to see if genistein has any effect on preventing or reducing heart disease and diabetes risk in men receiving Androgen Deprivation Therapy for prostate cancer. A combination of nutritional measures, blood markers and imaging tools will assess body composition, lipid levels and insulin resistance. Information from this pilot study will increase understanding of interventions which may prevent or reduce health risks during prostate cancer treatment. This project involves 24 men who will receive androgen deprivation therapy for prostate cancer.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled trial of daily oral genistein in 24 men initiating Androgen Deprivation Therapy (ADT) for prostate cancer (PCa). Genistein is a natural supplement that comes from soy. The purpose of this study is to see if genistein has any effect on preventing or reducing heart disease and diabetes risk in men receiving ADT for PCa. A combination of nutritional measures, blood markers and imaging tools will assess body composition, lipid levels and insulin resistance. Information from this study will increase understanding of interventions which may prevent or reduce health risks during prostate cancer treatment.

All participants will receive standard counseling for diet and exercise by their oncology care team. Participants will be asked to withhold from any additional dietary supplements (with the exception of 1 standard daily multivitamin) during the study period. Participants will also be asked to complete a food diary for three days (on two weekdays and 1 weekend day).

Subjects will be randomized and stratified by diabetes status to either 60 mg/day oral genistein (30 mg taken twice daily), or matching placebo. The goal for randomizing based on diabetes status is to ensure approximately the same number of subjects who have diabetes and do not have diabetes receive genistein and placebo.

During follow-up, subjects will receive weekly reminders via phone call, text, or email to enhance compliance and monitor for potential adverse events. The 3-month study visit will be scheduled to coincide with the subject's standard of care follow-up visit. Three-month assessments will be the same as baseline assessments.

Investigators seek to assess indexes of insulin dynamics (insulin sensitivity and secretion) determined from an oral glucose tolerance test before and 12 weeks after a daily genistein or placebo supplement. Measures of vascular function before and 12 weeks after a daily genistein or placebo supplement will also be assessed via ultrasound along with other metabolic measures via blood draw.

ELIGIBILITY:
Inclusion Criteria:

* Medical indication for androgen deprivation therapy (ADT) via luteinizing hormone-releasing hormone (LHRH) analog ± oral anti-androgen
* Diagnosis of prostate cancer
* ECOG performance status ≤ 2
* Life expectancy > 6 months
* Ability to provide informed consent

Exclusion Criteria:

* Transmural myocardial infarction, unstable angina, or congestive heart failure requiring hospitalization within the last 6 months
* Acute coronary event within the past month
* Use of intravenous antibiotics within the last 6 months
* Chronic liver disease
* Current use of cytotoxic or immunosuppressive drugs
* Chronic glucocorticoid or acute glucocorticoid or other synthetic steroid intake within the last month
* Chronic diarrhea or malabsorptive diseases (e.g., Crohn's disease)
* Stage 5 chronic kidney disease or need for hemodialysis
* Supplemental oxygen dependency
* Brain metastasis
* Severe cognitive dysfunction impairing ability to provide informed consent or consume study drug
* Dysphagia or requirement for artificial feeding
* Surgery or hospitalization within the last month
* Chemotherapy or radiation therapy within the last 60 days
* Insulin dependent diabetes
* HIV/AIDS
* History of organ transplant
* ECOG performance status > 2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Alvarez, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between October 2017 and March 2021. 10 participants consented to take part in the study and 2 withdrew at some point in the study. Results are presented on all data provided by all participants before withdrawal, where applicable.
Groups:
- Genistein: Participants with and without diabetes received 60 mg/day oral genistein (30 mg taken twice daily).
  Genistein: Genistein is a natural supplement that comes from soy. Genistein was taken orally (30 mg twice daily).
  Treatment was intended for 12 weeks but due to study termination treatment only lasted up to 8 weeks.
- Placebo: Participants with and without diabetes received placebo taken twice daily.
  Placebo: A placebo pill was taken orally.
  Treatment was intended for 12 weeks but due to study termination treatment only lasted up to 8 weeks.
Period: Overall Study
Arm/Group | Genistein | Placebo
Started | 6 | 4
Completed | 5 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genistein | Placebo | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (5.2) | 65.3 (13.0) | 67.7 (8.7)
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.5 [67.0 to 73.0] | 67.5 [55.5 to 75.0] | 69.5 [63.0 to 73.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Matsuda Index of Whole-Body Insulin Sensitivity at Baseline and Week 8 Post-baseline
Description: The Matsuda index is a measurement of insulin sensitivity from plasma glucose and insulin concentrations during the oral glucose tolerance test (OGTT).
  Insulin sensitivity was calculated at baseline and after 8 weeks with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. Higher values are reflective of better insulin sensitivity. This test is not used to clinically diagnose disease, and there is no accepted, standard cutoff to define impaired insulin sensitivity or insulin resistance based on this index.
Time Frame: Baseline, Week 8 post-baseline
Population: Number of patients included only subjects that were able to complete the outcome assessment in each visit.
Measure: Median (Inter-Quartile Range); unit: index
Arm/Group | Genistein | Placebo
Number analyzed (Participants) | 6 | 3
index
  Baseline | 4.4 [2.4 to 5.5] | 6.1 [3.9 to 13.5]
  8 weeks post-baseline: number analyzed (Participants) | 5 | 2
  8 weeks post-baseline | 4.1 [2.1 to 4.4] | 7.7 [5.0 to 10.3]

2. Primary Outcome: β-cell Insulin Secretion Capacity Assessed by the Insulinogenic Index at Baseline and Week 8 Post-baseline
Description: β-cell insulin secretion was determined from the OGTT. It is calculated as the ratio of the change in insulin values over the first 30 minutes of the OGTT and the change in glucose values over the first 30 minutes. Higher values are reflective of higher insulin secretion. This test is not used to clinically diagnose disease, and there is no accepted, standard cutoff to define impaired insulin secretion based on this index.
Time Frame: Baseline, Week 8 post-baseline
Population: Number of patients included only subjects that were able to complete the outcome assessment in each visit.
Measure: Median (Inter-Quartile Range); unit: index
Arm/Group | Genistein | Placebo
Number analyzed (Participants) | 6 | 3
index
  Baseline | 1.1 [0.5 to 3.3] | 0.7 [0.5 to 1.3]
  Week 8 post-baseline: number analyzed (Participants) | 5 | 2
  Week 8 post-baseline | 2.1 [0.7 to 2.5] | 1.4 [1.4 to 1.4]

3. Secondary Outcome: Arterial Stiffness
Description: Arterial stiffness will be assessed by applanation tonometry. Results will be reported in m/s (meters/seconds). A higher value indicates a worse outcome.
Time Frame: Baseline, Week 8
Population: Number of patients included only subjects that were able to complete the outcome assessment in each visit.
Measure: Median (Inter-Quartile Range); unit: m/s
Arm/Group | Genistein | Placebo
Number analyzed (Participants) | 6 | 3
m/s
  Baseline | 7.4 [6.1 to 9.2] | 7.2 [7.1 to 8.5]
  Week 8: number analyzed (Participants) | 5 | 3
  Week 8 | 9.1 [7.9 to 9.5] | 7.2 [6.0 to 8.6]

4. Secondary Outcome: Vascular Endothelial Function at Baseline and Week 8 Post-baseline
Description: Vascular endothelial function was measured with flow-mediated dilation (FMD in %) via ultrasound. A lower FMD indicates a worse outcome.
Time Frame: Baseline, Week 8 post-baseline
Population: Number of patients included only subjects that were able to complete the outcome assessment in each visit.
Measure: Median (Inter-Quartile Range); unit: percentage of FMD
Arm/Group | Genistein | Placebo
Number analyzed (Participants) | 6 | 4
percentage of FMD
  Baseline | 4.9 [3.4 to 5.2] | 4.7 [2.4 to 6.3]
  Week 8 post-baseline: number analyzed (Participants) | 5 | 3
  Week 8 post-baseline | 4.4 [2.0 to 6.6] | 2.7 [1.1 to 8.4]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored weekly throughout the 8 weeks that participants were enrolled in the study.
Description: AEs were defined as undesirable medical events or experiences, and classified as "expected", "unanticipated", or "serious" adverse events. Serious adverse events (SAEs) were predefined as experiences that suggest a significant hazard, such as events which: a) are fatal, b) are life-threatening, c) result in permanent disability, d) require inpatient hospitalization, or e) involve cancer, a congenital anomaly, or drug overdose.
Arm/Group | Genistein | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 5/6 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genistein (N=6) | Placebo (N=4)
Flu (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Localized edema in feet and ankles (General disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Heat strokes (General disorders) | 1 (1) | 0 (0)
Swollen ankles (General disorders) | 0 (0) | 1 (2)
Oral surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Left hip soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 1 (1)
Constipation and diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (2)
Bone infection (Osteomyelitis) (Infections and infestations) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rash - upper arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abdominal discomfort (General disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Hair loss on fingers (General disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)
Overheating (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT02766478/Prot_SAP_000.pdf